CLINICAL TRIAL: NCT06509139
Title: Optimal Treatment Duration of Bismuth Quadruple Therapy for Helicobacter Pylori Eradication in Female Patients and Comparison of the Efficacy with That of Male Patients
Brief Title: Optimal Duration of Bismuth Quadruple Therapy for Helicobacter Pylori Eradication in Females As Compared with Males
Status: Enrolling by invitation | Phase: Phase 4 | Type: Interventional
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: A-BR-113-029
Record Dates: First submitted 2024-06-17; First posted 2024-07-19 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-06

CONDITIONS: Helicobacter Pylori Infection; Sex; Bismuth Quadruple Therapy
MeSH Terms: conditions — Coitus | interventions — bismuth tripotassium dicitrate; Tablets; Esomeprazole; Metronidazole; Tetracycline

STUDY DESIGN:
Intervention Model Description: Among the H. pylori-infected female patients, they are randomized to the 14-day bismuth-based quadruple therapy group and the 10-day bismuth-based quadruple therapy group to receive a 14-day and 10-day course, respectively, of the bismuth-based quadruple therapy. Afterward, the patients stop taking the proton pump inhibitor and antibiotics for 4 to 6 weeks, and then they receive 13C-urea breath test or an H. pylori stool antigen test to confirm successful eradication or not.
  The study also investigates the efficacy of the 10-day bismuth quadruple therapy between females and males following the above interventional study model.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- The 10-day bismuth-based quadruple therapy group for females (Active Comparator): The female patients receive a 10-day course of the bismuth-based quadruple therapy, including esomeprazole (Nexium 40 mg) 1 tab twice a day, bismuth subcitrate (dibismuth trioxide) (KCB F.C. 120 mg) 1 tab four times a day, metronidazole (Fuliclin 250 mg) 2 tab thrice a day, and tetracycline (250 mg) 2 tab four times a day.
  Interventions: Drug: Drug: Bismuth Subcitrate 120 MG Oral Tablet; Drug: Esomeprazole 40mg; Drug: Metronidazole 250 MG; Drug: Tetracycline Pill
- The 14-day bismuth-based quadruple therapy group for females (Active Comparator): The female patients receive a 14-day course of the bismuth-based quadruple therapy, including esomeprazole (Nexium 40 mg) 1 tab twice a day, bismuth subcitrate (dibismuth trioxide) (KCB F.C. 120 mg) 1 tab four times a day, metronidazole (Fuliclin 250 mg) 2 tab thrice a day, and tetracycline (250 mg) 2 tab four times a day.
  Interventions: Drug: Drug: Bismuth Subcitrate 120 MG Oral Tablet; Drug: Esomeprazole 40mg; Drug: Metronidazole 250 MG; Drug: Tetracycline Pill
- The 10-day bismuth-based quadruple therapy group for males (Active Comparator): The male patients receive a 10-day course of the bismuth-based quadruple therapy, including esomeprazole (Nexium 40 mg) 1 tab twice a day, bismuth subcitrate (dibismuth trioxide) (KCB F.C. 120 mg) 1 tab four times a day, metronidazole (Fuliclin 250 mg) 2 tab thrice a day, and tetracycline (250 mg) 2 tab four times a day.
  Interventions: Drug: Drug: Bismuth Subcitrate 120 MG Oral Tablet; Drug: Esomeprazole 40mg; Drug: Metronidazole 250 MG; Drug: Tetracycline Pill

INTERVENTIONS:
Drug: Drug: Bismuth Subcitrate 120 MG Oral Tablet — Bismuth Subcitrate (120 MG Oral Tablet) 1 tab per oral four times per day for 14 days in the14-day bismuth-based quadruple therapy and for 10 days in the10-day bismuth-based quadruple therapy
  Other Names: KCB F.C.
Drug: Esomeprazole 40mg — Esomeprazole (40 mg) 1 tab per oral twice per day for 14 days in the14-day bismuth-based quadruple therapy and for 10 days in the10-day bismuth-based quadruple therapy
  Other Names: Nexium
Drug: Metronidazole 250 MG — Metronidazole (250 MG) 2 tab per oral thrice per day for 14 days in the14-day bismuth-based quadruple therapy and for 10 days in the10-day bismuth-based quadruple therapy
  Other Names: Fuliclin
Drug: Tetracycline Pill — Tetracycline (250 MG) 2 tab per oral four times per day for 14 days in the14-day bismuth-based quadruple therapy and for 10 days in the10-day bismuth-based quadruple therapy
  Other Names: Tetracycline (250 mg)

SUMMARY:
Helicobacter pylori eradication can reduce the risk of gastric cancer and decrease the recurrence of ulcers. However, in recent years, the increasing antibiotic resistance of Helicobacter pylori has reduced the efficacy of clarithromycin-based triple therapy to below 80%. The recent studies, including real-world data and a clinical trial, have consistently found that females have poorer eradication rate of Helicobacter pylori as compared with males. In previous clinical trial, investigators discovered that the efficacy of a 10-day bismuth quadruple therapy was not inferior to a 14-day bismuth quadruple therapy. However, it remains to be investigated whether the 10-day bismuth quadruple therapy is still non-inferior to the 14-day regimen in females.

This project continues the clinical trial to investigate whether the efficacy of the 10-day bismuth quadruple therapy in females is inferior to that in males and whether the 14-day bismuth quadruple therapy is superior to the 10-day regimen in females. The ultimate goal is to establish that male patients can use the 10-day bismuth quadruple therapy with fewer side effects and without compromising efficacy as compared with the 14-day regimen; while female patients are recommended to use the 14-day bismuth quadruple therapy as it would be more effective than the 10-day regimen.

Considering sex in research is becoming increasingly important, as females have more antibiotic-resistant Helicobacter pylori infection than males. The bismuth quadruple therapy can overcome most resistance issues. Researching and comparing the difference in the efficacy of bismuth quadruple therapy for Helicobacter pylori eradication between females and males are of significant clinical importance and align with current research trends.

DETAILED DESCRIPTION:
The recently published real-world study on Helicobacter pylori treatment, revealing that female (odds ratio 2.41 [95% confidence interval (CI) 1.16-5.03], P = 0.02) and age-Charlson Comorbidity Index ≥ 2 (odds ratio 3.16 [1.05-9.48], P = 0.04) were two independent factors for the failure of sequential therapy in eradicating Helicobacter pylori. The main cause of eradication failure is antibiotic resistance of the bacteria. Previous studies have found that females had more antibiotic-resistant Helicobacter pylori infections as compared with males did. In Australia and Italy, female was a predictor of metronidazole resistance; in Japan and Korea, female was a predictor of clarithromycin resistance; and among Alaskan Natives and in China, female predicted resistance to both metronidazole and clarithromycin.

The recent clinical trial found that the efficacy of a 10-day bismuth quadruple therapy was non-inferior to a 14-day bismuth quadruple therapy (Intention-to-treat analyses, 92.4% [95% (CI): 88.2%-96.5%] vs. 92.9% [95% CI: 88.9%-97.0%], absolute difference: -0.6%, lower boundary of the one-sided 97.5% CI: -6.7%, P = 0.020). However, subgroup analyses for males and females showed that while the 10-day therapy remained non-inferior to the 14-day therapy in males (95.2% [95% CI: 90.6%-99.8%] vs. 94.0% [95% CI: 88.4%-99.7%], absolute difference: 1.2%, lower boundary of the one-sided 97.5% CI: -6.8%, P = 0.022), it could not be demonstrated as non-inferior in females (89.2% [95% CI: 82.1%-96.3%] vs. 92.1% [95% CI: 86.5%-96.3%], absolute difference: -3.0%, lower boundary of the one-sided 97.5% CI: -12.3%, P = 0.198).

Previous research has identified female as a factor in the failure of 7-day clarithromycin-based triple therapy or concomitant therapy for Helicobacter pylori eradication. However, it is still uncertain whether female is a factor for Helicobacter pylori eradication failure with bismuth quadruple therapy.

In recent years, analyzing research results separately for females and males has become a trend. Historically, gender and sex differences were often overlooked in research design, conduct, and reporting, limiting the generalizability and applicability of findings to clinical practice. Heidari et al. have also advocated for the establishment of basic principles for international guidelines to encourage interdisciplinary research to systematically report sex and gender differences. The Sex and Gender Equity in Research (SAGER) guidelines recommend that researchers provide information on sex and gender in research design, data analysis, and result interpretation.

Given consecutive findings that females may have lower Helicobacter pylori eradication rates than males, designing a study to compare the efficacy of different durations of bismuth quadruple therapy between sexes is of significant clinical importance and aligns with current research trends.

This study hypothesizes that the rate of antibiotic resistance is higher in females compared to males. Consequently, the 10-day bismuth quadruple therapy will have a lower eradication rate in females compared to males. Because of the higher level of antibiotic resistance, females may require a longer treatment duration of 14 days to achieve the optimal eradication rate.

The patients with Helicobacter pylori infection are enrolled from National Cheng Kung University Hospital and Tainan Hospital, Ministry of Health and Welfare. Enrolled male participants received 10-day bismuth quadruple therapy. Enrolled female participants were randomly assigned into 10- or 14-day bismuth quadruple therapy with a 1:1 allocation ratio. Females and males are defined by biological attributes based on external body characteristics.

Sample size assessment: Using a Chi-square test to compare the 10-day bismuth quadruple therapy in females (experimental group) with the 10-day bismuth quadruple therapy in males (control group), where the efficacy in the control group is 96%. The null hypothesis is that there is no difference in efficacy between the experimental and control groups, with a margin of difference set at 7% (Helicobacter pylori eradication rate must be at least 90%). If the efficacy difference between the two groups is ≥ 7% (experimental group efficacy < 90%), the null hypothesis will be rejected, indicating a difference between females and males in efficacy of the 10-day bismuth quadruple therapy. If the efficacy difference between the two groups is < 7% (experimental group efficacy ≥ 90%), the null hypothesis cannot be rejected; however, there is no evidence to suggest that the 10-day therapy in females is as effective as in males. Based on this, each group needs 221 patients to achieve 80% power and a two-sided 95% confidence interval to reject the null hypothesis of a ≥ 7% difference in efficacy between the two groups.

Additionally, a superiority trial will compare the 14-day bismuth quadruple therapy in females (experimental group) with the 10-day bismuth quadruple therapy in females (control group), where the efficacy in the control group is 89%. The null hypothesis is that the experimental group is the same as or worse than the control group, with a margin of difference set at 7% (past research shows bismuth quadruple therapy efficacy at 96%). If the experimental group is superior to the control group with a difference of ≥ 7% (experimental group efficacy ≥ 96%), the null hypothesis will be rejected, indicating that the 14-day therapy is superior to the 10-day therapy in females. If the efficacy difference between the two groups is < 7% (experimental group efficacy < 96%), the null hypothesis cannot be rejected; however, there is no evidence to suggest that the 14-day therapy is as effective as or worse than the 10-day therapy in females. Based on this, each group needs 219 patients to achieve 80% power and a two-sided 95% confidence interval to reject the null hypothesis of a < 7% difference in efficacy between the two groups.

Primary Endpoint: The primary endpoint of the study is the successful eradication rate of Helicobacter pylori. All enrolled participants will be included in the overall analysis, incorporating intention-to-treat, per-protocol, and modified intention-to-treat analyses. All enrolled participants are included in the intention-to-treat analysis; those who are lost to follow-up, take less than 80% of the study medications, or have any protocol violation are excluded from the per-protocol analysis. The modified intention-to-treat analysis is similar to the intention-to-treat analysis, but patients with missing primary outcome data are excluded.

Secondary Endpoints: The secondary endpoints include the incidence of adverse events and medication adherence. There are 14 adverse events recorded, including dizziness, skin rash, headache, taste alteration, abdominal pain, nausea, diarrhea, constipation, bloating, vomiting, tongue discoloration, darkened stool, fatigue, and anorexia. Adverse events are assessed by a physician and a format questionnaire survey after the end of treatment. Serious adverse events are defined as daily activities restricted or participant unable to work. Medication adherence is assessed using a medication diary to record the number of days the medication was taken.

Statistical analysis: The statistical analysis is performed with SPSS software (SPSS 17, Chicago, IL, USA). The Student's t-test, Pearson's χ2 test, and Mann-Whitney U test are conducted to identify the statistical differences between the two comparison groups.

Antibiotic resistance that might affect the eradication rate, is assessed by H pylori culture.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are > 18 years
* H. pylori infection confirmed by histology of a gastric biopsy, a positive rapid urease test, or a positive 13C-urea breath test.

Exclusion Criteria:

* History of H. pylori eradication
* Previous allergic reactions to any drugs in the bismuth quadruple therapy
* Severe comorbidities
* Pregnant or breastfeeding women

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Females and males are defined by biological attributes based on external body characteristics
Enrollment: 661 (Estimated)
Dates: Start 2024-07-09 (Actual); Primary Completion 2032-07-31 (Estimated); Study Completion 2032-07-31 (Estimated)

PRIMARY OUTCOMES:
The successful eradication rate | About 4 to 6 weeks after receiving the H. pylori eradication regimen
  The patients stop taking the proton pump inhibitor and antibiotics for 4 to 6 weeks, and then they receive 13C-urea breath test or an H. pylori stool antigen test to confirm successful eradication or not. The successful rate is represented with a percentage (%).

SECONDARY OUTCOMES:
Adverse effects of the bismuth-based quadruple therapy | Since 1st day to 4 weeks after receiving the H. pylori eradication regimen
  Adverse event rates are assessed by physicians and through questionnaire surveys after treatment completion. Adverse events include dizziness, skin rash, headache, unpleasant taste, abdominal pain, nausea, vomiting, diarrhea, constipation, abdominal fullness, glossitis, darkened stool, fatigue, and anorexia. All adverse events are classified as none, mild (not restricting daily activities), or serious (restricting daily activities or causing inability to work).
Adherence to medications of the bismuth-based quadruple therapy | Since 1st day to 4 weeks after receiving the H. pylori eradication regimen
  Medication adherence is assessed by physicians and through questionnaire surveys after treatment completion. Medication adherence is categorized as good (≥ 80% medication taken) or poor (< 80% medication taken).

CONTACTS AND LOCATIONS:
Overall Officials: Hsiu-Chi Cheng, MD, PhD, Study Chair — Department of Internal Medicine, National Cheng Kung University Hospital, Tainan, Taiwan
Locations (1):
- Helicobacter pylori study group, National Cheng Kung University Hospital, Tainan, Taiwan

IPD SHARING:
Plan to Share IPD: No